CLINICAL TRIAL: NCT00493129
Title: ONTAK (Denileukin Diftitox) in Patients With Systemic Mastocytosis
Brief Title: Ontak (Denileukin Diftitox) in Patients With Systemic Mastocytosis (SM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0142
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Leukemia; Systemic Mastocytosis
Keywords: Systemic Mastocytosis; SM; Mast Cell Leukemia; Leukemia; Denileukin Diftitox; Ontak
MeSH Terms: conditions — Leukemia; Mastocytosis, Systemic; Leukemia, Mast-Cell | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ontak (Experimental): Ontak administered intravenously on Days 1-5 at the dose of 9 µg/kg/day, with a rest period from Days 6-21.
  Interventions: Drug: Ontak (Denileukin Diftitox)

INTERVENTIONS:
Drug: Ontak (Denileukin Diftitox) — 9 µg/kg by vein Days 1-5 of a 21 day cycle.
  Other Names: Denileukin Diftitox

SUMMARY:
Primary Objective:

1. To assess the response rate of ONTAK in Systemic Mastocytosis (SM) patients.

Secondary Objectives:

1. To assess the safety of ONTAK in SM patients.
2. To evaluate the time to progression and duration of response following treatment with ONTAK.

DETAILED DESCRIPTION:
Denileukin diftitox has been used for the treatment of a variety of disorders, in particular, malignant lymphoma, another blood-related disease. Denileukin diftitox is believed to be able to specifically attach to and kill malignant mast cells.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have blood (around 2 teaspoons) and bone marrow samples collected. To collect a bone marrow sample, an area of the hip bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. These samples will be used for tests to confirm the diagnosis of the disease. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible, you will receive denileukin diftitox as an injection by vein once a day for 5 days in a row. This will be repeated every 3 weeks (1 cycle). You will receive treatment on an outpatient basis. Treatment will continue as long as there is evidence that therapy is affecting the disease and is beneficial to you. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

During treatment you will have blood (around 1 teaspoon) collected twice during every 3-week period. You will also have bone marrow samples collected every 3 months during the treatment.

After the end of treatment, blood and bone marrow samples will be collected every 3 months until the disease gets worse or you start a different therapy. The blood and bone marrow samples will be used to look at response to therapy.

This is an investigational study. Denileukin diftitox has been approved by the FDA for the treatment of skin T-cell lymphoma and is commercially available. The use of denileukin diftitox in this study is investigational. You will be provided denileukin diftitox free of charge. Up to 25 participants will take part in this study. All be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SM, including mast cell leukemia (MCL).
* ECOG Performance Status (PS) 0-3
* Adequate renal function (indicated by serum creatinine </= 2.5 mg/dL); adequate hepatic function (indicated by ALT </= 3 * upper limit of normal; total bilirubin </= 3 * upper limit of normal; and albumin >/= 2.8 g/dL).
* Provide written informed consent.
* Female patients of childbearing potential must have a negative pregnancy test within 14 days prior to first dose of study drug, and must agree to use an effective means of contraception following the pregnancy test, throughout the study and for at least three weeks after their last treatment on protocol.

Exclusion Criteria:

* History of hypersensitivity to diphtheria toxin.
* Active cardiovascular disease as defined by New York Heart Association (NYHA) Class III-IV categorization.
* Serious intercurrent medical illnesses or active infections requiring parenteral antibiotics that would interfere with the ability of the patient to carry out the treatment program.
* Concurrent malignancy (other than resected basal or squamous cell skin cancers or in-situ cervical cancer). Unless, patient has SM-associated clonal hematologic disease that does not require therapy, as judged by treating physician and approved by principal investigator.
* Female patients who are pregnant or breastfeeding.
* No chemotherapy, radiotherapy, immunotherapy, hormonal anticancer therapy, or experimental medications (including approved drugs tested in an investigational setting) may be administered while a patient is a participant in this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 3 months
  Bone marrow samples used to look at response to therapy collected every 3 months until disease progression or different therapy started. Clinical efficacy assessed as objective response (major and partial response) for responding patients analyzed by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org